CLINICAL TRIAL: NCT02313597
Title: Outcomes in High Perianal Fistula Repair Using Video-assisted Anal Fistula Treatment Compared With Seton Use: a Randomized Controlled Trial
Brief Title: Video-assisted Anal Fistula Treatment Versus Seton in the Management of High Peri Anal Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. SamiUllah (Other Government)
Responsible Party: Sponsor-Investigator, Dr. SamiUllah, Medical Officer, Services Hospital, Lahore
Organization: Services Hospital, Lahore (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V1
Record Dates: First submitted 2014-08-28; First posted 2014-12-10 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Post Operative Pain; Recurrence
MeSH Terms: conditions — Pain, Postoperative; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SETON (Placebo Comparator): Silk suture will be used as SETON
  Interventions: Procedure: SETON
- VAAFT (Experimental): Video assisted anal fistula treatment
  Interventions: Procedure: VAAFT

INTERVENTIONS:
Procedure: SETON — In seton treatment, initially Hydrogen peroxide will be applied to the external opening with a 10-cc syringe, and the internal opening will be located by direct visualization of the anal canal via proctoscope. A probe will be inserted into the external opening and carefully maneuvered through the internal opening. Silk 1/0 suture will be then tied to the tip of the probe, which will be then squeezed out of the external opening. The suture will be then tied around the sphincter and through fistula tract. Later, the seton will be tightened at four-week intervals under local anesthesia until the suture cut through the sphincter.
  Arms: SETON
Procedure: VAAFT — Patients assigned to the VAAFT group will receive the following procedure. The external opening will be widened with a probe, and a fistulascope will be inserted to delineate the primary and secondary tracts and locate the internal opening. The internal opening will be then stitched with Vicryl™ (Polyglactin 910) 2-0 suture through the anal route with the help of a proctoscope. The tract of the fistula will be washed and debrided through the scope and cauterized. Finally, the external opening will be excised and will be sent for biopsy.
  Arms: VAAFT

SUMMARY:
Anal fistula is the most common Peri anal disease. It's a disease with an incidence of 9 in 100,000. Anal fistula is classified on the basis of its location into high and low anal fistula, above or below dentate line respectively.

Multiple series have shown that the formation of a fistula tract following anorectal abscess occurs in 7-40% of cases. There are typically 8-10 anal crypt glands at the level of the dentate line in the anal canal arranged circumstantially. These glands afford a path for infecting organisms to reach the intramuscular spaces. The cryptoglandular hypothesis states that an infection begins in the anal canal glands and progresses into the muscular wall of the anal sphincters to cause an anorectal abscess.

According to internal opening many author proposed certain classification but the standardized in all of them is Park's classification, so this study categorized the patient through this classification. There are four types of fistula-in-ano in Park's Classification intersphincteric (between internal and external sphincters is 70%), transsphincteric (across external sphincters is 25%), suprasphincteric (over sphincters), and extrasphincteric(above and through levator ani).High anal fistula is considered to be difficult to treat because of its location.This study diagnosed the internal opening of high perianal with the help of endoluminal ultrasound and MRI.

Classic method of its treatment are fistulotomy, fistulectomy and Setone placement but these are associated with lots of complication like fecal incontinence,recurrence,pain.Therefore many method have been recently devised including Ligation of intersphincteric fistula tract (Lift), glue repair and flap advancement.Another recently introduced method for its treatment is Video-assisted anal fistula treatment (VAAFT) proposed by P. Meinero which has been associated with less complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either gender with age ranging from 15 to 60 years.
2. All patients with high anal fistula

Exclusion Criteria:

1. Patients with suspected malignancy determined by the presence of a mass on digital rectal examination,
2. History of previous perianal surgery,
3. History of irritable bowel disease determined by medical record
4. Uncontrolled diabetes

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmood Ayyaz, FCPS FACS, Study Director — Professor of Surgery
Locations (1):
- Hospitals, Lahore, Punjab Province, Pakistan

RESULTS

PARTICIPANT FLOW:
Groups:
- SETON: Hydrogen peroxide was injected to the external opening with a 10-cc syringe, and the internal opening was located by direct visualization of the anal canal via proctoscope. A cannulating probe was inserted into the external opening and carefully maneuvered through the internal opening. Silk 1/0 suture was then tied to the tip of the probe, which was then squeezed out of the external opening. The suture was then tied around the sphincter and through fistula tract, Later, the seton was tightened at four week interval under spinal anesthesia until the suture cut through the sphincter.
- VAAFT: The external opening was widened with a probe, and a fistulascope was inserted to delineate the primary and secondary tracts and locate the internal opening. The internal opening was then stitched with Vicryl™(Polyglactin 910) 2-0 suture through the anal route with the help of a proctoscope. And the tract of the fistula was washed and debrided through scope and it was coagulated with cautry so that tract be closed.
Period: Overall Study
Arm/Group | SETON | VAAFT
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SETON | VAAFT | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.4 (10.1) | 39.9 (12.4) | 39.1 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 9 | 7 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Pakistan | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence of Disease or Fistula
Description: Number of Participants with Recurrence of Disease or Fistula 3 Years After Treatment
Time Frame: 3 years postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | SETON | VAAFT
Number analyzed (Participants) | 40 | 40
Participants | 5 | 10

2. Secondary Outcome: Duration of Surgery
Description: Duration of surgery measured upto 180 minutes
Time Frame: Time from beginning of surgery to end of surgery,assessed up to 180 minutes
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | SETON | VAAFT
Number analyzed (Participants) | 40 | 40
Minutes | 36.97 (12.98) | 78.60 (26.24)

3. Secondary Outcome: Pain Score
Description: Pain score measured through visual analog score with 1 being minimum and 10 being maximum. Lesser value represents better outcome and greater value shows worse outcome.
Time Frame: 12 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SETON | VAAFT
Number analyzed (Participants) | 40 | 40
score on a scale | 2.82 (1.58) | 4.22 (1.83)

4. Secondary Outcome: Time to Return to Work
Time Frame: up to 4 weeks
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | SETON | VAAFT
Number analyzed (Participants) | 40 | 40
Days | 9.27 (2.06) | 7.42 (1.78)

5. Secondary Outcome: Time to Healing of Fistula
Time Frame: up to 12 weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | SETON | VAAFT
Number analyzed (Participants) | 40 | 40
weeks | 9.7 (1.87) | 5.75 (1.17)

ADVERSE EVENTS:
Time Frame: up to 12 weeks
Arm/Group | SETON | VAAFT
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
One of the limitations of our study is that it is single center study and results cannot be generalized, another thing is that we did not inject glue after doing VAAFT into remaining tract (as advised by Monre who is the inventor of this procedure) and we do not know whether this injection of glue can affect recurrence of fistula or not.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT02313597/Prot_SAP_000.pdf